CLINICAL TRIAL: NCT05634746
Title: Fluticasone Propionate Oral Disintegrating Tablet Formulation in Eosinophilic Esophagitis: A Randomized, Double-blind, Placebo-Controlled 24-Week Induction Study of APT-1011, Followed by a Single-arm Open-label Extension, in Adult Subjects With Eosinophilic Esophagitis
Brief Title: 24-Week Induction Study of APT-1011 in Adult Subjects With Eosinophilic Esophagitis (EoE) (FLUTE 3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ellodi Pharmaceuticals, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-1011-005
Expanded Access: NCT05095116 (No longer available)
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Eosinophilic Esophagitis
Keywords: APT-1011; Esophagitis; Eosinophilic Esophagitis; Esophageal Diseases; Gastrointestinal Diseases; Digestive System Diseases; Gastroenteritis; Eosinophilia; Leukocyte Disorders; Hematologic Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases; Fluticasone; Anti-Inflammatory Agents; Bronchodilator Agents; Autonomic Agents; Peripheral Nervous System Agents; Anti-Asthmatic Agents; Respiratory System Agents; Anti-Allergic Agents; FLUTE 3; FLUTE III; Flute
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis; Esophageal Diseases; Gastrointestinal Diseases; Digestive System Diseases; Gastroenteritis; Eosinophilia; Leukocyte Disorders; Hematologic Diseases; Hypersensitivity, Immediate; Hypersensitivity; Immune System Diseases | interventions — APT-1011; Endoscopy, Digestive System

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- APT-1011 (Experimental): APT-1011 3 mg HS
  Interventions: Drug: APT-1011; Procedure: Esophagogastroduodenoscopy
- Placebo (Placebo Comparator): Placebo HS
  Interventions: Drug: Placebo oral tablet; Procedure: Esophagogastroduodenoscopy

INTERVENTIONS:
Drug: APT-1011 — APT-1011 is an orally disintegrating tablet that includes fluticasone propionate as its active ingredient.
  Other Names:
  fluticasone propionate
  Arms: APT-1011
Drug: Placebo oral tablet — Placebo orally disintegrating tablet.
  Other Names:
  PBO
  Arms: Placebo
Procedure: Esophagogastroduodenoscopy — Esophagogastroduodenoscopy (EGD) is a test that involves an endoscope, a lighted camera on the end of a tube, that is passed down a subject's throat to visualize their esophagus

SUMMARY:
This is a 24-week randomized, double-blind, placebo-controlled induction study of APT-1011 in adults (≥18 years old) with eosinophilic esophagitis (EoE) followed by a single-arm, open-label extension. This study will evaluate the efficacy and safety of APT-1011 3 mg administered HS (hora somni, at bedtime) for the induction of response to treatment (symptomatic and histologic) over 24 weeks. The open-label extension will continue to evaluate long-term safety in subjects who consent to continue on open-label treatment with APT-1011.

DETAILED DESCRIPTION:
The efficacy and safety of APT-1011 3 mg administered at bedtime will be evaluated for the induction of response (histologic and symptomatic) after 24 weeks of treatment. After completing 24 weeks of double-blind study treatment, subjects may consent to participate in the open-label extension, otherwise they will complete study drug treatment and enter a 2-week off treatment safety follow-up.

The duration of the double-blind portion of the study, screening through follow-up visit for subjects completing study drug at Week 24, will be up to 32 weeks long, i.e., 6-week screening period (the includes a 4-week run-in phase) followed by 24 weeks induction phase and 2 weeks off-treatment follow-up. For subjects consenting to participate in the open-label extension, the duration of the study will be determined by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female ≥18 years of age at the time of informed consent
2. Each subject must read, understand, and provide consent on the ICF for this study and be willing and able to adhere to study-related treatment regimens, procedures, and visit schedule
3. Diagnosis or presumptive diagnosis of EoE that is confirmed during the Screening period by histology that demonstrates ≥15 peak eos/HPF. In order to ensure that a diagnosis can be made, at least 6 biopsies should be taken in total from both proximal and distal esophageal mucosal areas (at least 3 each). Mid-esophageal biopsies are not required (optional). HPF will be defined as a standard area of 235 square microns in a microscope with 40x lens (0.3 mm^2) and 22 mm ocular.

   1. Esophagogastroduodenoscopies and biopsies are to be obtained during the Screening period
   2. Biopsies will be read by a central pathologist
   3. Esophagogastroduodenoscopies and biopsies performed outside the study will not be accepted to meet eligibility criteria
   4. Optional biopsies may be taken and processed locally for local use, only where specified in the local ICF. If serious pathology is unexpectedly encountered biopsies of such lesions must be processed locally
4. Have a subject-reported history of ≥6 episodes to a maximum of 30 episodes of dysphagia in a 14-consecutive-day period within 18 days prior to baseline
5. Completion of the evening eDiary on at least 11 out of the 14-consecutive-day observation period during the 4-week run-in period (Baseline Symptom Assessment).The minimum requirement of 11 days need not be consecutive.

Exclusion Criteria:

1. Have known contraindication, hypersensitivity, or intolerance to corticosteroids
2. Have a contraindication to, or factors that substantially increase the risk of, EGD procedure or esophageal biopsy or have narrowing of the esophagus that precludes EGD with a standard (8-10 mm) endoscope
3. Have history of an esophageal stricture requiring dilatation within the 12 weeks prior to Screening
4. Have any physical, mental, or social condition or history of illness or laboratory abnormality that in the Investigator's judgment might interfere with study procedures or the ability of the subject to adhere to and complete the study or increase the safety risk to the subject such as uncontrolled diabetes or hypertension
5. History of recurrent or current oral or esophageal mucosal infection due to inhaled or nasal corticosteroids
6. Have any mouth or dental condition that prevents normal eating (excluding braces)
7. Have any condition affecting the esophageal mucosa or altering esophageal motility other than EoE, including erosive esophagitis (grade B or higher as per the Los Angeles Classification of Gastroesophageal Reflux Disease; hiatus hernia longer than 3 cm, Barrett's esophagus, and achalasia)
8. Use of systemic (oral or parenteral) corticosteroids within 30 days before Screening, use of swallowed corticosteroids within 30 days before Screening
9. Initiation of either inhaled or nasal corticosteroids or high-potency dermal topical corticosteroids within 30 days before Screening
10. Use of calcineurin inhibitors or purine analogues (azathioprine, 6-mercaptopurine) in the 12 weeks before Screening
11. Use of potent cytochrome P450 (CYP) 3A4 inhibitors (e.g., ritonavir and ketoconazole) in the 4 weeks before Screening
12. Initiation of an elimination diet or elemental diet within 30 days before Screening (diet must remain stable after signing ICF)
13. Abnormal ACTH stimulation defined as a serum cortisol level <16 μg/dL (440 nmol/L) at 60 minutes with ACTH stimulation test using 250 μg cosyntropin
14. Use of biologic immunomodulators, including dupilumab for EoE, with dose last administered within 6 months before Screening (allergy desensitization injection or oral therapies allowed as long as the course of therapy is not altered during the study period)
15. Subjects who have initiated, discontinued, or changed dosage regimen of histamine H2 receptor antagonists, antacids or antihistamines, leukotriene inhibitors, or sodium cromolyn within 4 weeks before qualifying endoscopy during Screening. If already receiving these drugs, the dosage must remain constant throughout the study
16. Subjects who have initiated PPIs within 8 weeks before qualifying endoscopy. If already receiving PPIs, the dosage regimen must remain constant throughout the study
17. Have gastrointestinal bleeding or documented active peptic ulcer within 4 weeks prior to Screening or entering a new study period
18. Have chronic infection such as prior or active tuberculosis, active chicken pox or measles, or absence of prior measles, mumps, and rubella vaccine. Subjects with tuberculosis exposure or who live in, or travel to, high endemic areas should be assessed locally for tuberculosis before consideration for the study
19. Immunosuppression or immunodeficiency disorder
20. Current malignancy or malignancy within 3 years of Screening, with the exception of skin cancers other than melanoma. Subjects in remission for at least 3 years post-treatment may be enrolled.
21. Have a history or presence of Crohn's disease, celiac disease, or other inflammatory disease of the gastrointestinal tract, including non-EoE eosinophilic gastrointestinal disorders (EGIDs)
22. Have current drug abuse in the opinion of the Investigator
23. Have current alcohol abuse in the opinion of the Investigator
24. Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study
25. Sexually active females of childbearing potential who do not agree to follow highly effective contraceptive methods through the End of Study visit
26. Have received an investigational product as part of a clinical trial within 30 days (or 5 half-lives, whichever is longest) of Screening. Subjects who are currently participating in observational studies or enrolled in patient registries are allowed in this study
27. Have participated in a prior study with investigational product APT-1011

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Histological Remission (Co-Primary Outcome Measure) | Week 24
  To evaluate the percentage of subjects with histological remission (defined ≤ 6 peak eosinophils [eos]/high power field [HPF] on esophageal mucosal biopsies at Week 24). HPF will be defined as a standard area of 235 square microns in a microscope with 40x lens (0.3 mm^2) and 22 mm ocular
Complete Symptomatic Response (Co-Primary Outcome Measure) | Week 24
  To evaluate the percentage of subjects with complete symptomatic response at Week 24 (defined as zero dysphagia episodes in the 14 consecutive days prior to Week 24)

SECONDARY OUTCOMES:
Clinicopathologic Responder Rate | Week 24
  To compare the percentage of clinicopathologic responders, defined as having complete symptomatic AND histological response at Week 24 (defined as zero dysphagia episodes in the 14 consecutive days prior to Week 24 AND ≤ 6 peak eos/HPF on esophageal mucosal biopsies)
Percentage of Subjects with ≥70% Reduction in Dysphagia Frequency | Week 24
  To evaluate the percentage of subjects with ≥70% reduction in dysphagia frequency at Week 24 as compared to baseline (as measured over the 14 consecutive days prior to each visit)
Mean Change in Dysphagia Frequency | Week 24
  To compare the mean change from baseline to Week 24 in dysphagia frequency (as measured over the 14 consecutive days prior to each visit)
Mean Change in PROSE Difficulty Swallowing | Week 24
  To compare the mean change from baseline to Week 24 in difficulty swallowing using the Patient Reported Outcomes Symptoms of Eosinophilic Esophagitis (PROSE)
Mean Change in PROSE Pain with Swallowing | Week 24
  To compare the mean change from baseline to Week 24 in pain with swallowing using the PROSE
Mean Number of Dysphagia-Free Days | Week 24
  To compare the mean number of dysphagia-free days from baseline to Week 24
Percentage of Responders (Strictures and ≥Grade 2 rings) | Week 24
  To compare the percentage of responders, defined as no longer having strictures and/or ≥Grade 2 rings which were present at baseline, at Week 24
Percentage of Responders (Strictures) | Week 24
  To compare the percentage of responders, defined as no longer having strictures which were present at baseline, at Week 24
Percentage of Responders (≥Grade 2 rings) | Week 24
  To compare the percentage of responders, defined as no longer having ≥Grade 2 rings which were present at baseline, at Week 24
Mean Change in EREFs | Week 24
  To compare endoscopic appearance evaluated by the mean change from baseline to Week 24 in Eosinophilic Esophagitis Endoscopic Reference Score (EREFs)
Time to First Complete Symptom Response | Week 24
  Time to first complete symptom response (defined as zero dysphagia episodes in a 14-consecutive-day period)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Dellon, MD, MPH, Principal Investigator — UNC Center for Esophageal Diseases and Swallowing
Locations (60):
- United States (59):
  - Digestive Health Specialists, Dothan, Alabama
  - East View Medical Research LLC, Mobile, Alabama
  - Premier Allergy Asthma and Immunology, Scottsdale, Arizona
  - Del Sol Research Management, LLC., Tucson, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Om Research LLC, Camarillo, California
  - Providence Facey Medical Foundation, Mission Hills, California
  - United Medical Doctors, Murrieta, California
  - TriWest Research Associates, LLC, San Diego, California
  - Precision Research Institute, LLC, San Diego, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Western States Clinical Research, Inc., Wheat Ridge, Colorado
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Nature Coast Clinical Research, Inverness, Florida
  - I.H.S Health, LLC, Kissimmee, Florida
  - Endoscopic Research Inc, Orlando, Florida
  - Revival Clinical Research, Orlando, Florida
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - GI Alliance - Glenview, Glenview, Illinois
  - GI Alliance - Gurnee, Gurnee, Illinois
  - Deaconess Clinic Allergy, Evansville, Indiana
  - Gastroenterology Health Partners, PLLC, New Albany, Indiana
  - Velocity Clinical Research, Inc., Overland Park, Kansas
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Gastro Center of Maryland, LLC, Columbia, Maryland
  - Velocity Clinical Research, Inc., Rockville, Maryland
  - Boston Specialists, Boston, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Henry Ford Health System, Novi, Michigan
  - Clinical Research Institute of Michigan, LLC, Troy, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - MNGI Digestive Health, P.A., Plymouth, Minnesota
  - Clinical Research Professionals, Chesterfield, Missouri
  - Bozeman Health, Bozeman, Montana
  - Advanced Research Institute, Reno, Nevada
  - New Mexico Clinical Research & Osteoporosis Center, Inc., Albuquerque, New Mexico
  - New York Gastroenterology Associates, New York, New York
  - UNC Clinical and Translational Research Center (CTRC), Chapel Hill, North Carolina
  - Charlotte Gastroenterology & Hepatology, PLLC, Charlotte, North Carolina
  - Carolina Research, Greenville, North Carolina
  - Bernstein Clinical Research, Cincinnati, Ohio
  - Centricity Research Columbus, Columbus, Ohio
  - Northshore Gastroenterology Research, LLC, Westlake, Ohio
  - Vital Prospects Clinical Research Institute., PC, Tulsa, Oklahoma
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC, Uniontown, Pennsylvania
  - Rapid City Medical Center, LLP, Rapid City, South Dakota
  - Texas Digestive Specialists, Harlingen, Texas
  - GI Alliance, Lubbock, Texas
  - GI Alliance, Mansfield, Texas
  - Southern Star Research Institute, LLC., San Antonio, Texas
  - GI Alliance, Webster, Texas
  - Advanced Research Institute, Ogden, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Advanced Research Institute, Sandy City, Utah
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Washington Gastroenterology, PLLC dba GI Alliance, Bellevue, Washington
  - GI Alliance, Tacoma, Washington
- Joel Liem Medicine Professional Corporation, Windsor, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No